CLINICAL TRIAL: NCT02190149
Title: Study of Prophylaxis, ACtivity and Effectiveness (SPACE) in Hemophilia Patients Currently Treated With ADVATE or RIXUBIS
Acronym: SPACE
Status: Completed | Type: Observational
Sponsor: Baxalta now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Other Study IDs: 061302
Record Dates: First submitted 2014-07-14; First posted 2014-07-15 (Estimated); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Hemophilia A; Hemophilia B
Keywords: Factor VIII Deficiency; Factor FIX Deficiency
MeSH Terms: conditions — Hemophilia A; Hemophilia B | interventions — Factor VIII; F8 protein, human; Factor IX

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ADVATE (Factor VIII): Participants will remain on their current (pre-study) treatment regimen of ADVATE throughout the study period
  Interventions: Biological: ADVATE (Antihemophilic Factor [Recombinant])
- RIXUBIS (Factor IX): Participants will remain on their current (pre-study) treatment regimen of RIXUBIS throughout the study period
  Interventions: Biological: RIXUBIS (Coagulation Factor IX [Recombinant])

INTERVENTIONS:
Biological: ADVATE (Antihemophilic Factor [Recombinant])
  Other Names: Octocog alfa
  Groups: ADVATE (Factor VIII)
Biological: RIXUBIS (Coagulation Factor IX [Recombinant])
  Groups: RIXUBIS (Factor IX)

SUMMARY:
This 6-month prospective outcomes study addresses the association between timing of infusion, patient activity levels, and bleeding episodes through patient-reported measurements.

ELIGIBILITY:
Inclusion Criteria:

* 13 to 65 years old at the time of screening
* has moderately severe or severe hemophilia A or B (FVIII/FIX level

  ≤2%), with or without transient inhibitors
* Hemophilia A patient currently prescribed ADVATE (FVIII) or Hemophilia B patient currently prescribed RIXUBIS (FIX)
* previously treated with plasma-derived FVIII/FIX concentrates or recombinant FVIII/FIX for ≥150 documented exposure days (EDs)
* is willing and able to comply with the requirements of the protocol
* is proficient in the English language to allow for use of the SPACE eDiary

Exclusion Criteria:

* inhibitor titer ≥0.6 Bethesda units or currently being treated for an inhibitor
* has participated in another clinical study involving a medicinal product or device within 30 days prior to enrollment or is scheduled to participate in another clinical study involving a medicinal product or device during the course of this study
* is a family member or employee of the investigator
* elective major surgery is planned within 6 months after enrollment which may interfere with activities of daily living (at investigator's discretion)
* continuously require walking assistance devices (eg, wheelchair, crutches, etc.)

Ages: 13 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hemophilia treatment center (HTCs) in the US will be identified and invited to enroll eligible patients in this study
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2014-07-22 (Actual); Primary Completion 2016-03-29 (Actual); Study Completion 2016-03-29 (Actual)

PRIMARY OUTCOMES:
Advancing the understanding of the relationship between patient physical activity levels, infusion and occurrence of bleeding episodes (BEs) | 6 months retrospectively (after the informed consent form (ICF) is signed) through 6 months
  After the informed consent form is signed, retrospective data on physical activity levels, infusion and occurrence of BEs will be collected. The retrospective period will be the 6 months prior to signing the ICF.

SECONDARY OUTCOMES:
Types of current physical activities of participants | Baseline through 6 months
Activity measurement | Baseline through 6 months
  Including: calories burned, steps taken, distance traveled, and active minutes
Infusion schedule for participants on prophylaxis | Baseline through 6 months
Infusion amount (either ADVATE (Hemophilia A), or RIXUBIS (Hemophilia B) | Baseline through 6 months
Occurrence of bleeding episodes (BEs) | 6 months retrospectively (after the informed consent form (ICF) is signed) through 6 months
  After the informed consent form is signed, retrospective data on physical activity levels, infusion and occurrence of BEs will be collected. The retrospective period will be the 6 months prior to signing the ICF.
Patient-reported outcome: Hemophilia Activities List (HAL) questionnaire - for adult patients | Baseline and 6 months
  The HAL measures activities involving the upper extremities, basic activities involving the lower extremities and complex activities involving the lower extremities as well as an overall physical activity score for adults.
Patient-reported outcome: pediatric Hemophilia Activities List (pedHAL) questionnaire - for pediatric patients | Baseline and 6 months
  The PedHAL measures activities involving the upper extremities, basic activities involving the lower extremities and complex activities involving the lower extremities as well as an overall physical activity score for participants 13-17 years of age:

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (17):
- United States (17):
  - Orthopaedic Hospital DBA Orthopaedic Hemophilia Treatment Center, Los Angeles, California
  - Rady Childrens Hospital, San Diego, California
  - University of Colorado, Aurora, Colorado
  - Bleeding and Clotting Disorders Institute, Peoria, Illinois
  - University of Kentucky Medical Center, Lexington, Kentucky
  - Johns Hopkins University School Of Medicine, Baltimore, Maryland
  - Childrens Hospital of Michigan, Detroit, Michigan
  - Michigan State University, East Lansing, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Children's Mercy Hospitals & Clinics, Kansas City, Missouri
  - North Shore/Long Island Jewish PRIME, Great Neck, New York
  - The Presbyterian Hospital, Charlotte, North Carolina
  - Oregon Health & Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - The Vanderbilt Clinic, Nashville, Tennessee
  - The University of Texas MD Anderson, Harlingen, Texas
  - Puget Sound Blood Center, Seattle, Washington

REFERENCES:
- See also: To obtain more information on the study, click here/on this link. — https://clinicaltrials.takeda.com/study-detail/5f6b5fc24db2bf003ab457fd